CLINICAL TRIAL: NCT06442917
Title: The Effect of Breathing Exercise and Affirmation Method Used in Labor on Women's Birth Self-Efficacy and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Collaborators: Mehmet Akif Ersoy Canakkale State Hospital (Other Government)
Responsible Party: Principal Investigator, Remziye Gültepe, PhD, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20.478.486/1213
Record Dates: First submitted 2024-05-22; First posted 2024-06-04 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Birth Self-efficacy; Birth Satisfaction
Keywords: self-efficacy; self-satisfaction; breathing exercise; affirmation
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breathing Exercise Group (Experimental): 32 the Pregnant Identifying Characteristics Form, the Short Version of the Self-Efficacy Scale in Childbirth was completed before the pregnancy intervention and the VAS was measured.
  Interventions: Behavioral: Breathing Exercise
- Affirmation Method Group (Experimental): 32 pregnant women who were admitted to the hospital for childbirth and were in the latent phase (0-3 cm) filled out the pre-intervention Pregnant Identifying Characteristics Form, the Short Version of the Self-Efficacy Scale in Childbirth, and the VAS was measured.
  Interventions: Behavioral: Affirmation Method
- Breathing Exercise and Affirmation Method Group (Experimental): During the latent phase, affirmation phrases were shown to the pregnant women and the application was explained and the application was made with breathing exercise training.
  Interventions: Behavioral: Breathing Exercise and Affirmation Method
- control group (No Intervention): Routine midwifery care was applied during the trauma.

INTERVENTIONS:
Behavioral: Breathing Exercise — 32 the Pregnant Identifying Characteristics Form, the Short Version of the Self-Efficacy Scale in Childbirth was completed before the pregnancy intervention and the VAS was measured. Breathing exercise training and application were carried out during the latent phase process. In this training, the importance of proper breathing was explained and diaphragmatic breathing application was made.
  During the active phase process (4-7 cm), the Innatal Period Evaluation Form was filled out and the VAS was measured, and diaphragmatic breathing exercise was performed every 30 minutes from the beginning of contraction until the end of contraction. During the transition phase (8-10 cm), the Innatal Period Evaluation Form, the Short Version of the Self-Efficacy Scale in Childbirth were filled out and the VAS was measured, and diaphragmatic breathing exercise was performed once every 15 minutes from the beginning of contraction to the end of contraction.
  Arms: Breathing Exercise Group
Behavioral: Affirmation Method — 32 pregnant women who were admitted to the hospital for childbirth and were in the latent phase (0-3 cm) filled out the pre-intervention Pregnant Identifying Characteristics Form, the Short Version of the Self-Efficacy Scale in Childbirth, and the VAS was measured. During the latent phase, affirmation phrases were shown to the pregnant women and the application was explained. During the active phase process (4-7 cm), the Innatal Period Evaluation Form was filled out and the VAS was measured, and the affirmation phrases were repeated and used by the researcher every 30 minutes from the beginning of the contraction until the end of the contraction.
  During the transition phase (8-10 cm), the Innatal Period Evaluation Form, the Short Version of the Self-Efficacy Scale in Childbirth were filled out and the VAS was measured, and affirmation sentences and support sentences were said every 15 minutes from the beginning of the contraction to the end of the contraction.
  Arms: Affirmation Method Group
Behavioral: Breathing Exercise and Affirmation Method — During the latent phase, affirmation phrases were shown to the pregnant women and the application was explained and the application was made with breathing exercise training. In this training, the importance of proper breathing was explained and diaphragmatic breathing application was made. During the active phase process (4-7 cm), the Congenital Period Evaluation Form was filled out and the VAS was measured, and diaphragmatic breathing exercise was performed once every 30 minutes from the beginning of contraction to the end of contraction, and the affirmation phrases were repeated and used by the researcher
  Arms: Breathing Exercise and Affirmation Method Group

SUMMARY:
Purpose: This research was conducted to determine the effect of breathing exercise and affirmation method used in labor on women's birth self-efficacy and satisfaction.

Materials and Methods: The sample of the study, in which the randomized controlled experimental design type was applied, consisted of 128 nulliparous pregnant women. Data were collected with Pregnant Descriptive Information Form, Innate Period Evaluation Form, Visual Analog Scale, Affirmation Statement Evaluation Form, Short Form of the Childbirth of Self-Efficacy Inventory and Birth Satisfaction Scale. Pregnant women who are in the first stage of labor have been using diaphragmatic breathing exercise to one group, affirmation method to one group, both diaphragmatic exercise and affirmation method to one group since the active phase, while pregnant women in the control group have not been given any intervention, they have received routine care. Descriptive statistical methods, chi-square test, one-way analysis of variance, t-test for dependent and independent groups were used in the analysis of the data.

DETAILED DESCRIPTION:
This study was conducted in four groups. Groups; The group in which the affirmation method was used in labor (Affirmation Group - OG), the group in which breathing exercises were used in labor (Breathing Group - NG), the group in which both breathing exercises and affirmation methods were used in labor (Breathing and Affirmation Group - NOG), and the group in which no intervention was made other than routine hospital practices. It is divided into a non-existent group (Control Group - CG). The numbers given to the groups (1, 2, 3, 4) were determined by the lottery method. The name of each group was written on the papers and numbered in order of drawing. The numbers 3 were assigned to the Breathing group, 1 to the Affirmation group, 2 to the Breathing and Affirmation group, and 4 to the Control group. Considering data loss in the distribution of the study into groups, numbers from 1 to 200 were randomized for 4 groups using a computer-assisted randomization program (https://www.rstudio.com). In order to ensure homogeneity in the randomization of the intervention groups and the control group, five matching criteria were taken into consideration. These match criteria; It was determined as the mother's age, education level (secondary school and below, high school and above), employment status (working/not working), gestational age, and prenatal education. Homogeneity of the groups was tested in the evaluation of the study.

Pregnant women to be included in the study were assigned to groups according to the numbers in the columns according to the eligibility criteria. In order to avoid being influenced by each other, pregnant women were included in the study one by one, and after the birth of one pregnant woman was completed, the other pregnant woman was included in the study.

ELIGIBILITY:
Inclusion Criteria:

The one who is open to communication,

* between the ages of 18-45 Dec,
* At least a primary school graduate,

  * Nulliparous,
* Non-risky pregnancy in terms of mother and baby (multiple pregnancy, preeclampsia, etc.),

  * In the first stage of labor (0-3 cm dilatation), which is,
* Living at term and having a single pregnancy,
* No analgesic or anesthetic substance is applied during the trauma, * Pregnant women who volunteer to participate in the research

Exclusion Criteria:

* Your mother wants to leave without working, * Pregnant women who developed cesarean section indication after being included in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Woman
Enrollment: 128 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
birth self-efficacy scale | in the active phase of labor
  birth self-efficacy of pregnant women.The lowest total score that can be obtained from the scale is 32, and the highest total score is 320. As the scores from the scale increase, the self-efficacy levels of pregnant women in labor increase.
birth satisfaction scale | in the active phase of labor
  birth satisfaction of pregnant women.As a result of the scale, a score between 0 and 40 is received. It is interpreted that as the score obtained as a result of the scale increases, the woman's birth satisfaction increases, while a low score indicates that the birth satisfaction is not at a sufficient level.

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart Üniversitesi, Çanakkale, Turkey (Türkiye)